CLINICAL TRIAL: NCT07019545
Title: A PHASE II TRIAL AIMING TO INVESTIGATE THE SAFETY AND CLINICAL ACTIVITY OF BELANTAMAB MAFODOTIN IN ADULT PATIENTS WITH PRIMARY IMMUNE THROMBOCYTOPENIA PREVIOUSLY TREATED WITH A THROMBOPOIETIN RECEPTOR AGONIST AND/OR RITUXIMAB AFTER CORTICOSTEROID FIRST-LINE THERAPY
Acronym: BONSAI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Society of Hematology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EAE140; 2023-509131-12-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — belantamab mafodotin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): Trial treatment is defined as the combination of belantamab mafodotin plus dexamethasone. Trial treatment is given in 28-day cycles for a total period of one year per patient or until treatment failure (loss of response), physician decision, unacceptable toxicity, withdrawal of consent, or death (whichever occurs first). Participants without confirmed response or better after two infusions with belantamab mafodotin, and the interval following the dosing, will be discontinued from trial treatment and will not be replaced.
  Interventions: Drug: Belantamab Mafodotin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Belantamab Mafodotin — Belantamab mafodotin is administered intravenously (IV) at a dose of 1.9 mg/kg on Day 1 of every other 28-day cycle for the first two administrations and then 1.9 mg/kg on Day 1 of every third 28-day cycle.
Drug: Dexamethasone — Dexamethasone is administered IV or per OS (PO) at a dose of 40 mg/day on days 1, 2, 3, 4 and 15, 16, 17, 18 of every 28-day cycle for the first two cycles in participants <75 years; at 20 mg/day on days 1, 2, 3, 4 and 15, 16, 17, 18 of every 28-day cycle for the first two cycles in participants ≥75 years.

SUMMARY:
This is a Phase II open label, prospective, multicenter trial designed to assess the safety and clinical activity of belantamab mafodotin in adult patients with primary immune thrombocytopenia (ITP) previously treated with a thrombopoietin receptor agonist (TPO-RA) and/or rituximab after first-line treatment with corticosteroids. Overall, 14 participants will be enrolled in the trial. Participants' follow-up will continue for up to 12 months after the last participant is enrolled. The accrual period will be approximately 12 months.

Trial treatment will be given in 28-day cycles for a total period of one year per patient or until treatment failure, physician decision, unacceptable toxicity, withdrawal of consent, or death (whichever occurs first). Participants without confirmed Response (R) or better after two infusions with belantamab mafodotin will be discontinued from trial treatment and will not be replaced.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 years or older.
2. Primary ITP with platelet cell count of less than 30x10^9/L.
3. Prior first-line therapy with corticosteroids.
4. Prior second-line therapy with TPO-RA and/or rituximab and failure to achieve or retain response.
5. Adequate organ system function as defined by the below laboratory assessments. Hematologic

   1. Absolute neutrophil count ≥1.5 X 10^9/L; granulocyte colony stimulating factor use within the past 14 days is NOT permitted.
   2. Hemoglobin ≥8.0 g/dL; transfusions within the past 14 days are NOT permitted. Erythropoietin use is allowed. Hepatic

   <!-- -->

   1. Total bilirubin ≤1.5xULN (isolated bilirubin ≥1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
   2. Alanine aminotransferase ≤ 2.5xULN. Renal

   a. Estimate glomerular filtration rate ≥30 mL/min/1.73 m^2; calculated using the Modified Diet in Renal Disease formula.
6. Female participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical trials: A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

   * Is not a woman of childbearing potential (WOCBP) defined as follows:

     1. ≥45 years of age and has not had menses for >1 year.
     2. Participants who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation.
     3. Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure. OR
   * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency during the intervention period and for 4 months after the last dose of belantamab mafodotin and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of trial intervention.
   * WOCBP must have a negative highly sensitive serum pregnancy test at screening within 72 hours of dosing on C1D1 and agree to use a highly effective method of contraception during the trial and for 4 months after the last dose of belantamab mafodotin. Additional requirements for pregnancy testing during and after trial intervention are provided in Section 10. Trial Procedures and Visit Schedule. The investigator is responsible for a review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with a nearly undetected pregnancy.
7. Male participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical trials: Male participants are eligible to participate if they agree to the following during the intervention period and until 6 months after the last dose of belantamab mafodotin, whichever is longer, to allow for clearance of any altered sperm.

   • Refrain from donating sperm

   PLUS either:
   * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent, OR
   * Must agree to use contraception/barrier as detailed below:

   Agree to use a male condom, even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year as when having sexual intercourse with a woman of childbearing potential (including pregnant females).
8. Eastern Cooperative Oncology Group Performance (ECOG) Status ≤ 2.
9. Participants must be able to understand the trial procedures and agree to participate in the trial by providing written informed consent.

Exclusion Criteria:

1. Secondary ITP including:

   i. Drug induced ITP. ii. ITP associated with any autoimmune disorders (e.g., systemic lupus erythematosus and rheumatoid arthritis). iii. ITP associated with chronic infection (e.g., human immunodeficiency virus, hepatitis C virus and helicobacter pylori). iv. ITP associated with malignancy (e.g., chronic lymphocytic leukemia or large granular T-lymphocyte lymphocytic leukemia). v. ITP associated with chronic infection.
2. Chronic liver disease. Cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, persistent jaundice. NOTE: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) is acceptable if participant otherwise meets entry criteria.
3. To be seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]) at screening or within 3 months prior to first dose of trial treatment.

   NOTE 1: Participants with resolved infection (i.e., participants who are positive for antibodies to hepatitis B core antigen [anti-HBc] or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR). Those who are PCR positive will be excluded.

   NOTE 2: presence of ant-iHBs indicating previous vaccination will not constitute an exclusion criterion.
4. To be seropositive for hepatitis C at screening or within 3 months prior to first dose of trial treatment.

   NOTE: Participants with positive hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained. Hepatitis RNA testing is optional and participants with negative hepatitis C antibody test are not required to also undergo hepatitis C RNA testing.
5. Known HIV infection unless the participant can meet all of the following criteria:

   1. Established anti-retroviral therapy (ART) for at least 4 weeks and HIV viral load <400 copies/mL
   2. CD4+ T-cell (CD4+) counts ≥350 cells/uL
   3. No history of AIDS-defining opportunistic infections within the last 12 months NOTE: consideration must be given to ART and prophylactic antimicrobials that may have a drug:drug interaction and/or overlapping toxicities with belantamab mafodotin or other combination products as relevant.
6. Active infection requiring treatment.
7. Presence of active renal condition (infection, requirement for dialysis, or any other significant condition that could affect participant's safety).
8. Any serious and/or unstable pre-existing medical or psychiatric disorder, or other conditions (including laboratory abnormalities) that could interfere with participant's safety, obtaining informed consent, or compliance to the trial procedures.
9. Participant must not have received a live or live-attenuated vaccine within 30 days prior to first dose of belantamab mafodotin.
10. Current corneal epithelial disease except for mild punctate keratopathy. NOTE: Participants with mild punctate keratopathy are allowed. Mild (Grade 1) punctuate keratopathy is characterized by the appearance of only a few, if any, microcyst-like epithelial changes, as identified in the slit-lamp examination, with a low density (non-confluent), and predominantly (≥80%) located in the periphery of the cornea.
11. Known intolerance or immediate or delayed hypersensitivity reaction or idiosyncratic reaction to: drugs chemically related to belantamab mafodotin, or any of the components of the trial treatment; or infused protein products, sucrose, histidine, and polysorbate 80.
12. Use of an investigational drug within 14 days or 5 half-lives (whichever is shorter) preceding the first dose of trial drug.
13. Prior treatment with a monoclonal antibody within 30 days of receiving the first dose of trial drug. Please note, monoclonal antibodies for serious conditions unrelated to MM, such as COVID, may be permitted but need to be discussed with the Sponsor.
14. Symptomatic amyloidosis, active POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal plasmaproliferative disorder, skin changes) or active plasma cell leukemia at the time of screening.
15. Evidence of active mucosal or internal bleeding.
16. Ongoing Grade 2 or higher peripheral neuropathy or neuropathic pain.
17. Major surgery within 4 weeks before the first dose of trial drug NOTE 1: participant must be clinically stable following a major surgery to be entered in the trial.

NOTE 2: major surgery shall be defined based on the Investigator's judgment according to the extent and complexity of the procedure, its pathophysiological consequences and consecutive clinical outcomes. 18. Evidence of cardiovascular risk including any of the following: i. Evidence of current clinically significant untreated arrhythmias, including clinically significant ECG abnormalities, second degree (Mobitz Type II), or third degree atrioventricular block. ii. Screening 12-lead ECG showing a baseline QT interval >470 msec iii. History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 3 months of Screening. iv. Class III or IV heart failure as defined by the New York Heart Association functional classification system (Appendix 3 - New York Heart association (NYHA) Classification v. Uncontrolled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy of treatment with belantamab mafodotin in terms of Complete response rate (CRR)/Partial response rate (PRR) | At 6 months of treatment
  CRR/PRR is defined as the percentage of participants with a confirmed best response of PR or CR (Response-evaluable population). The denominator will be the total number of participants in the Response-evaluable population.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Athens "Alexandra", Athens, Attica, Athens, Greece

IPD SHARING:
Plan to Share IPD: No